CLINICAL TRIAL: NCT01218828
Title: Hydration With Different Sodium Chloride Protocols for the Prevention of Contrast Medium-induced Nephropathy in Patients Undergoing Coronary Angiography: a Randomized Trial
Brief Title: Prevention of Contrast Renal Injury With Different Hydration Strategies
Acronym: POSEIDON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KP-RCCL-5718
Record Dates: First submitted 2010-10-08; First posted 2010-10-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Contrast Medium-induced Nephropathy
Keywords: Contrast; nephropathy; cardiac catheterization; angiography; percutaneous coronary intervention is
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard therapy (Active Comparator): Hydration with 0.9% saline per a standard protocol (control group)
  Interventions: Other: Standard hydration
- LVEDP-based hydration strategy (Experimental): LVEDP guided hydration with 0.9% saline (treatment group)
  Interventions: Other: LVEDP -Based hydration strategy

INTERVENTIONS:
Other: LVEDP -Based hydration strategy
  Arms: LVEDP-based hydration strategy
Other: Standard hydration
  Arms: Standard therapy

SUMMARY:
Using a randomized controlled trial design, two hydration protocols for the prevention of contrast medium-induced nephropathy will be tested.

DETAILED DESCRIPTION:
The study population will be recruited from subjects undergoing cardiac catheterization.

Subjects will be randomized to one of two hydration protocols:

1. normal saline at 3 mL/kg for one hour prior to contrast exposure and 1.5 mL/kg/hr during and for four hours post procedure.
2. normal saline at 3 mL/kg for one hour prior to contrast exposure and then the fluid rate would be adjusted according to the left ventricular end diastolic pressure (LVEDP). The fluid rate based upon the LVEDP measurement is maintained during the procedure and for four hours post procedure. The LVEDP hydration strategy follows: (2A) < 13 mmHg, 5 mL/kg/hr during and for four hours post procedure. (2B) 13-18 mmHg, 3 mL/kg during and for four hours post procedure. (2C) > 18 mmHg, 1.5 mL/kg during and four hours post procedure.

Renal function assessment will be made using standard laboratory measures post procedure.

ELIGIBILITY:
Inclusion Criteria:

* estimated GFR less than or equal to 60 mL/min/1.73 m^2
* age greater than 18 years
* at least one of the following: diabetes mellitus, history of congestive heart failure, hypertension, or age greater than 75 years.

Exclusion Criteria:

* patients unable to give consent
* undergoing emergency cardiac catheterization
* on renal replacement therapy
* exposure to contrast media within the prior two days
* pulmonary edema or active congestive heart failure
* kidney transplant status
* severe valvular abnormalities
* change in serum creatinine greater than 15% over the prior two days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2010-10; Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Contrast induced nephropathy | Within four days of contrast exposure

SECONDARY OUTCOMES:
Renal replacement therapy, myocardial infarction, all-cause mortality | 30 days and long-term

CONTACTS AND LOCATIONS:
Overall Officials: Somjot S Brar, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, Los Angeles, California, United States

REFERENCES:
- [Derived] Brar SS, Aharonian V, Mansukhani P, Moore N, Shen AY, Jorgensen M, Dua A, Short L, Kane K. Haemodynamic-guided fluid administration for the prevention of contrast-induced acute kidney injury: the POSEIDON randomised controlled trial. Lancet. 2014 May 24;383(9931):1814-23. doi: 10.1016/S0140-6736(14)60689-9. PMID 24856027